CLINICAL TRIAL: NCT07393490
Title: The Effect of Apneic Oxygenation of the Non-ventilated Lung on the Expression of Hypoxia-inducible Factor-1 Alpha (HIF-1α) and Interleukin-6 (IL-6) in Lung Tissue During Lung Cancer Surgery.
Brief Title: Effect of Apneic Oxygenation of the Non-ventilated Lung During Lung Cancer Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APOXOS
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: One-lung ventilation; Apneic oxygenation; Inflammatory response; Hif 1 alpha; Interleukin 6; Thoracic anaesthesia
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Participants are assigned in parallel to either apneic oxygenation or standard ventilation during lung cancer surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apneic Oxygenation (Experimental): Patients receive apneic oxygenation of non-ventilated lung during lung cancer surgery.
  Interventions: Procedure: Apnoeic Oxygenation
- Control Group (Active Comparator): Patients receive standard ventilation during lung cancer surgery.
  Interventions: Procedure: Standard Ventilation

INTERVENTIONS:
Procedure: Apnoeic Oxygenation — Apneic oxygenation of the non-ventilated lung is applied during lung cancer surgery to maintain oxygenation and decrease inflammatory response while the lung is not mechanically ventilated.
  Arms: Apneic Oxygenation
Procedure: Standard Ventilation — Standard ventilation is applied during lung cancer surgery according to routine clinical practice.
  Arms: Control Group

SUMMARY:
This study investigates the effect of apneic oxygenation of the non-ventilated lung on local and systemic inflammatory response during lung cancer surgery.

Patients undergoing surgical resection of lung cancer often require one-lung ventilation during anaesthesia. This results in alveolar hypoxia accompanied by upregulated expression of inflammatory markers. Apneic oxygenation of the non-ventiladed lung may influence inflammatory processes and oxygenation during surgery. The aim of this study is to evaluate whether apneic oxygenation affects inflammatory markers in lung tissue and postoperative recovery in patients undergoing lung cancer surgery. The study is conducted at a single center and includes adult patients scheduled for elective lung cancer surgery. Data will be collected durig the perioperative period. The results of this study may contribute to improved anaesthetic management and patient outcomes during thoracic surgery.

DETAILED DESCRIPTION:
PARTICIPANTS:

This study will include 56 patients undergoing surgical lung resection for lung cancer. The patients will be divided into two groups: patients who will receive apneic oxygenation of the non-ventilated lung during surgery and patients who will not receive apneic oxygenation during lung resection for lung cancer.

MATERIALS AND METHODS

Preoperative Preparation and Randomization

All patients will undergo a preoperative evaluation prior to surgery, during which perioperative risk will be assessed based on existing comorbidities in accordance with the standardized protocol of the American Society of Anesthesiologists (ASA). Before surgery, and after providing written informed consent, baseline demographic data will be recorded, including age, sex, body weight, height, and body mass index (BMI). The presence of comorbidities and details of chronic medications will also be documented.

Patients will be randomized into two groups according to the use of intraoperative apneic oxygenation: patients in whom apneic oxygenation will be applied (AO group) and patients in whom apneic oxygenation will not be applied (control group, CO). Randomization will be performed using a computer-generated random number sequence with block randomization. The randomization process will be conducted by an independent individual. Allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes, which will be opened after patient enrollment in the study.

Prior to the start of surgery, blood samples will be collected from all participants for laboratory analysis, including complete blood count (CBC), differential blood count, C-reactive protein (CRP), procalcitonin (PCT), arterial blood gas analysis, and lactate levels.

Anesthesia and Surgical Procedure

Following preoxygenation via face mask (FiO₂ 1.0, flow rate 6 L/min, duration of four minutes), each patient enrolled in the study will receive induction of anesthesia with propofol (Propofol 1% MCT Fresenius, Fresenius Kabi, Bad Homburg, Germany) at a dose of 2 mg/kg, sufentanil (Sufentanyl Janssen, Janssen-Cilag, Beerse, Belgium) at a dose of 0.3 µg/kg, and rocuronium (Esmeron, NV Organon, Amsterdam, The Netherlands) at a dose of 0.6 mg/kg. A double-lumen endotracheal tube will be inserted to allow lung separation. Correct tube positioning will be confirmed by fiberoptic bronchoscopy (Ambu, Ballerup, Denmark).

Anesthesia will be maintained with continuous propofol infusion titrated according to bispectral index (BIS) values (Bispectral Index, Aspect Medical Systems Inc., Norwood, MA, USA), with additional administration of sufentanil and rocuronium based on clinical indicators and vital parameters.

In the apneic oxygenation (AO) group, a catheter will be placed under fiberoptic bronchoscopic guidance into the main bronchus of the isolated lung and connected to a separate breathing circuit delivering oxygen at a flow rate of 5 L/min; no such intervention will be performed in the control (CO) group. Immediately after thoracotomy, the surgeon will obtain a lung tissue sample from the non-ventilated lobe containing the tumor and scheduled for resection. The tissue sample will be used for immunohistochemical analysis at the Department of Pathology.

The non-operated lung will be ventilated using pressure-controlled ventilation, adjusted according to end-tidal CO₂ values (35-45 mmHg) and peripheral oxygen saturation (SpO₂ maintained > 90%). After resection of the lung lobe, an additional tissue sample will be collected for immunohistochemical processing and analysis of HIF-1α and IL-6 expression.

After completion of the surgery, patients will be awakened, extubated, and transferred to the intensive care unit for postoperative monitoring.

Intensive Care Unit Stay

During the first 24 hours of treatment in the intensive care unit, vital parameters will be continuously monitored and recorded hourly, including blood pressure, heart rate, peripheral oxygen saturation (SpO₂), body temperature, and urine output. On the day of surgery, six hours after completion of the surgical procedure, routine laboratory tests will be performed, including a complete blood count (CBC), as well as arterial blood gas analysis.

All patients will receive postoperative analgesic therapy consisting of paracetamol (Paracetamol, B. Braun, Melsungen, Germany) at a dose of 1 g every six hours and tramadol (Tramal, Stada Arzneimittel AG, Bad Vilbel, Germany) at a dose of 100 mg every six hours. Between these dosing intervals, patients will assess their pain, and in cases of breakthrough pain, meperidine (Dolsin, Pharma, Prague, Czech Republic) will be administered in 20 mg boluses. Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS), on which patients will rate their pain on a scale from 0 to 10, where 0 indicates no pain and 10 represents the worst imaginable pain.

Twenty-four hours after surgery, an additional set of laboratory tests will be performed, including complete blood count (CBC), differential blood count, C-reactive protein (CRP), procalcitonin (PCT), arterial blood gas analysis, and lactate levels.

Hospital Stay

During hospitalization, recovery of pulmonary function will be assessed daily based on the duration of postoperative oxygen therapy. Oxygen therapy will be discontinued once arterial oxygen partial pressure exceeds 8 kPa while breathing room air. While patients are receiving oxygen therapy, the oxygen flow rate delivered via face mask (in liters per minute) will be recorded.

For each patient, the total duration of stay in the intensive care unit, the overall length of hospital stay, the occurrence of all postoperative complications (including wound infection, postoperative bleeding, the need for reoperation, and adverse cardiovascular events), and the final treatment outcome-survival or death-will be documented.

Preparation of Specimens for Immunohistochemical Analysis

Lung tissue specimens obtained during surgery will be fixed in 10% buffered formalin (Biognost, Zagreb, Croatia) and processed using a Tissue-Tek VIP 6 automated tissue processor (Sakura Finetek, Tokyo, Japan). The specimens will then be embedded in paraffin blocks and sectioned at a thickness of 5 µm using a LEICA SM201R microtome (Leica Biosystems, Nussloch, Germany). Immunohistochemical analysis will be performed on a fully automated Ventana BenchMark Ultra platform (Roche, Basel, Switzerland).

Paraffin-embedded sections will be stained using antibodies against interleukin-6 (IL-6) and hypoxia-inducible factor-1 alpha (HIF-1α) (Abcam, Cambridge, UK).

Immunohistochemical Analysis

Histopathological analysis will be performed primarily in the alveolar regions of the lung parenchyma. Depending on the pathologist's assessment and the availability of representative tissue, examination of the bronchi, bronchioles, and interstitium may also be included. The expression of IL-6 and HIF-1α will be analyzed in three cellular compartments: inflammatory cells, vascular endothelial cells, and pneumocytes (alveolar epithelial cells).

For each sample, an area measuring 5 × 5 mm (25 mm²) will be analyzed. During area selection, regions with necrosis, collapsed or bullous alveolar spaces, folding artifacts, thickened section edges, or other structures that may hinder interpretation will be avoided. If a single section does not contain sufficient tissue to form one continuous area of 25 mm², several adjacent segments from the same sample will be analyzed, with a total analyzed area of 25 mm².

In each sample, the total number of positively stained cells will be counted for each cellular population. Positivity for IL-6 will be defined as cytoplasmic staining, whereas positivity for HIF-1α expression will be defined exclusively by nuclear staining. In addition, staining intensity will be recorded for each parameter using the following scale: 0 - no staining, 1 - weak staining, 2 - moderate staining, and 3 - strong staining.

The following controls will be included in each staining series: a positive control consisting of tissue sections with known physiological low-level expression of the target marker (breast carcinoma tissue for HIF-1α and appendix tissue with inflammatory cells for IL-6), a negative control achieved by omission of the primary antibody, and assessment of background staining as a visual control for nonspecific tissue staining.

Ethical Aspects of the Study

The study will involve physicians from the Department of Anesthesiology, Reanimatology and Intensive Care Medicine, the Department of Thoracic Surgery, and the Department of Pathology and Forensic Medicine of the University Hospital Center Osijek. The study will not alter the standard course of patient treatment in any way nor will it affect the quality of patient care.

All ethical principles outlined in relevant international, European, and national guidelines will be strictly adhered to throughout the study, in accordance with the Code of Ethics and Deontology of the Croatian Medical Association (2002), the Code of Ethics and Deontology of the Croatian Medical Chamber (2002), and other applicable international ethical documents.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients scheduled to undergo surgical resection of a single lung segment for lung cancer
* Written informed consent provided

Exclusion Criteria:

* Age younger than 18 years
* Chronic corticosteroid therapy and/or other immunomodulatory treatments
* Severe pulmonary diseases, including:

Chronic obstructive pulmonary disease classified as GOLD stage 3-4 (Global Initiative for Chronic Obstructive Lung Disease).

Severe asthma according to GINA classification (Global Initiative for Asthma), step 4.

Severe interstitial lung disease defined by: Forced vital capacity (FVC) < 50% predicted, diffusing capacity of the lung for carbon monoxide (DLCO) < 40% predicted, presence of extensive pulmonary fibrosis on computed tomography (CT)

* Surgical procedure expected to last less than 2 hours
* Intraoperative hemodynamic instability, defined as: Mean arterial pressure < 60 mmHg for more than 30 minutes despite adequate volume resuscitation, requirement for high-dose vasopressor support (norepinephrine > 0.2 µg/kg/min)
* New-onset intraoperative cardiac arrhythmias
* Significant intraoperative blood loss, defined as the need for transfusion of more than two units of packed red blood cells
* Intraoperative ventilatory instability, defined as: Severe hypoxemia (PaO₂ < 60 mmHg or SpO₂ < 85% with FiO₂ 1.0), hypercapnia (PaCO₂ > 70 mmHg with pH < 7.2), inability to achieve adequate ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Expression of HIF -1α in lung tissue | Intraoperative (during lung cancer surgery)
  Expression of hypoxia inducible factor 1 alpha (HIF 1α ) in lung tissue will be assessed to evaluate tissue hypoxia in patients receiving apneic oxygenation of the non-ventilated lung compared with those receiving standard ventilation during lung cancer surgery.
Expression of IL-6 in lung tissue | Intraoperative (during lung cancer surgery)
  Expression of interleukin 6 (IL-6) in lung tissue will be assessed to evaluate the local inflammatory response in patients receiving apneic oxygenation of the non-ventilated lung compared with those receiving standard ventilation during lung cancer surgery.

SECONDARY OUTCOMES:
Changes in leukocyte count | From preoperative baseline to 24 hours after surgery.
  Changes in peripheral blood leukocyte count from preoperative baseline will be measured to assess systemic inflammatory response associated with apneic oxygenation compared with standard ventilation.
Changes in neutrophile count | From preoperative baseline to 24 hours after surgery.
  Changes in peripheral blood neutrophil count from preoperative baseline will be measured to asses systemic inflammatory response associated with apneic oxygenation compared with standard ventilation.
Changes in arterial oxygen partial pressure (PaO2) | From preoperative baseline to 24 hours after surgery.
  Changes in arterial oxygen partial pressure (PaO2) from preoperative baseline will be measured to assess respiratory effects associated with apneic oxygenation compared with standard ventilation.
Changes in arterial carbon dioxide partial pressure (PaCO2) | From preoperative baseline to 24 hours after surgery.
  Changes in arterial carbon dioxide partial pressure (PaCO2) will be measured to assess respiratory effects associated with apneic oxygenation compared with standard ventilation.
Incidence of postoperative complications | Perioperative
  The incidence of postoperative complications occuring during the postoperative hospital stay will be recorded and compared between patients receiving apneic oxygenation and those receiving standard ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.